CLINICAL TRIAL: NCT03083886
Title: Spine Pain INtervention to Enhance Care Quality And Reduce Expenditure - Randomized Clinical Trial
Brief Title: Spine Pain INtervention to Enhance Care Quality And Reduce Expenditure
Acronym: SPINE CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Niteesh K. Choudhry, MD, PhD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017P000622
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Results first posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Back Pain; Neck Pain
MeSH Terms: conditions — Back Pain; Neck Pain | interventions — Ice; adenylate isopentenyltransferase

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual PCP led care (Active Comparator)
  Interventions: Other: Usual PCP led care
- Identify, Coordinated, Enhanced (ICE) Decision Making (Experimental)
  Interventions: Other: Identify, Coordinated, Enhanced (ICE) Decision Making + PCP led care
- Individualized Postural Therapy (IPT) (Experimental)
  Interventions: Other: Individualized Postural Therapy (IPT) + PCP led care

INTERVENTIONS:
Other: Identify, Coordinated, Enhanced (ICE) Decision Making + PCP led care — Subjects seeking care at a clinic assigned to this arm will receive the ICE care model through referral by their primary care provider. The ICE care model was developed by the Clinical Excellence Research Center at Stanford University based on a review of the peer-reviewed literature for adult subjects with incident neck or back pain less than six weeks in duration who are not using high-dose opioid medications or receiving spine-related long-term disability payments.
  Arms: Identify, Coordinated, Enhanced (ICE) Decision Making
Other: Individualized Postural Therapy (IPT) + PCP led care — IPT involves the evaluation of a subject's posture to identify postural and alignment deviations and, based on this, a personalized corrective exercise program is prescribed. This method does involve the use of prescription medications, surgery, or manipulation. A treatment course typically lasts eight sessions over eight weeks. In order to allow for the consistent delivery of this arm of the study at multiple study-sites across the country, IPT will be delivered by The Egoscue Method. Egoscue was founded in 1971 and has 25 clinics worldwide.
  Arms: Individualized Postural Therapy (IPT)
Other: Usual PCP led care — Primary care provider will direct patients' care pathway.
  Arms: Usual PCP led care

SUMMARY:
Low back and neck pain are among the leading causes of medical visits, lost productivity and disability. There is an urgent need to identify effective and efficient ways of helping subjects with acute spine pain while guiding practitioners towards high-value care. This trial will be a block and cluster-randomized open-label multi-centered pragmatic randomized clinical trial comparing healthcare spending and clinical outcomes for subjects with spine pain of less than three months' duration, in whom there are no red flag signs or symptoms. Subjects will be randomized to one of three treatment strategies: (1) usual primary care provider-led care; (2) usual PCP-led care with spine pain treatment directed by the Identify, Coordinate, and Enhanced decision making (ICE) care model, and (3) usual PCP-led care with spine pain treatment directed by the Individualized Postural Therapy (IPT) care model. Our outcomes of interest will be spine-related healthcare utilization at one year as well as pain and functionality of the study participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients with back or neck pain of ≤ 3 months' duration. All patients must have spine pain with or without radiation to the extremities or the head
* Age ≥ 18 years
* Willing and able to provide informed consent

Exclusion Criteria:

* Patients with symptoms attributed to the spine but without actual pain in the spine (e.g. those with cervicogenic headache without neck pain)
* Currently pregnant
* Currently receiving disability benefits, worker's compensation, or involved in litigation for a workplace injury
* Currently enrolled in another intervention trial for the management of acute back or neck pain
* Cancer that is metastatic or being actively treated. (i.e chemotherapy, radiation, surgery)
* History of receiving active therapy for back or neck pain in the past 3 months (7+ consecutive days of narcotic use, 6+ sessions of PT, chiropractic care, acupuncture, postural therapy, or other spine therapy delivered by a trained provider)
* History of spine surgery or spine injections/ablation in the past 6 months
* Severe, active psychosis or major depression inhibiting ability to physically participate in intervention
* Red Flag Symptoms (fever, night sweats, unintentional weight loss, bowel or bladder dysfunction, neurologic weakness, history of intravenous drug use)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3087 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niteesh K Choudhry, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (8):
- United States (8):
  - HonorHealth Medical Group, Phoenix, Arizona
  - Marwan A. Edris, MD, Laguna Hills, California
  - Teresa S. Sligh, MD, North Hollywood, California
  - Augusto Focil, MD, Oxnard, California
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Carlos R. Herrera, MD, Houston, Texas
  - Luis Zepeda, MD, Houston, Texas
  - Bernadette U. Iguh, MD, Houston, Texas

REFERENCES:
- [Derived] Choudhry NK, Fifer S, Fontanet CP, Archer KR, Sears E, Bhatkhande G, Haff N, Ghazinouri R, Coronado RA, Schneider BJ, Butterworth SW, Deogun H, Cooper A, Hsu E, Block S, Davidson CA, Shackelford CE, Goyal P, Milstein A; SPINE CARE Investigators; Crum K, Scott J, Marton K, Silva FM, Obeidalla S, Robinette PE, Lorenzana-DeWitt M, Bair CA, Sadun HJ, Goldfield N, Hogewood LM, Sterling EK, Pickney C, Koltun-Baker EJ, Swehla A, Ravikumar V, Malhotra S, Finney ST, Holliday L, Moolman KC, Coleman-Dockery S, Patel IB, Angel FB, Green JK, Mitchell K, McBean MR, Ghaffar M, Ermini SR, Carr AL, MacDonald J. Effect of a Biopsychosocial Intervention or Postural Therapy on Disability and Health Care Spending Among Patients With Acute and Subacute Spine Pain: The SPINE CARE Randomized Clinical Trial. JAMA. 2022 Dec 20;328(23):2334-2344. doi: 10.1001/jama.2022.22625. PMID 36538309
- [Derived] Choudhry NK, Fontanet CP, Ghazinouri R, Fifer S, Archer KR, Haff N, Butterworth SW, Deogun H, Block S, Cooper A, Sears E, Goyal P, Coronado RA, Schneider BJ, Hsu E, Milstein A. Design of the Spine Pain Intervention to Enhance Care Quality And Reduce Expenditure Trial (SPINE CARE) study: Methods and lessons from a multi-site pragmatic cluster randomized controlled trial. Contemp Clin Trials. 2021 Dec;111:106602. doi: 10.1016/j.cct.2021.106602. Epub 2021 Oct 22. PMID 34688915

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals ≥18 years with neck and/or back pain of ≤3 months' duration were eligible if they presented to one of the 33 participating primary care clinics in the U.S. between June 2017 and March 2020.
Pre-assignment Details: This study was randomized at the clinic level. Once clinics were randomized, all patients within that clinic were in that clinic's assigned arm. Patients who consented AND completed baseline questionnaires are included in the primary analytic dataset.
Units Other Than Participants: Clinics
Period: Overall Study
Arm/Group | Usual PCP Led Care | Identify, Coordinated, Enhanced (ICE) Decision Making | Individualized Postural Therapy (IPT)
Started (Patients who consented and enrolled) | 1035; 11 Clinics | 871; 11 Clinics | 1181; 11 Clinics
Completed Baseline Data (Patients who consented, enrolled, and provided baseline data. This is the primary analytic cohort.) | 992; 11 Clinics | 829; 11 Clinics | 1150; 11 Clinics
Completed | 940; 11 Clinics | 750; 11 Clinics | 1043; 11 Clinics
Not Completed | 95; 0 Clinics | 121; 0 Clinics | 138; 0 Clinics
Not completed — Withdrawal by Subject | 51 | 73 | 104
Not completed — Missing Baseline data | 43 | 42 | 31
Not completed — Investigator terminated | 1 | 6 | 3

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all patients who consented AND completed baseline questionnaires. This is the primary analytic cohort.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual PCP Led Care | Identify, Coordinated, Enhanced (ICE) Decision Making | Individualized Postural Therapy (IPT) | Total
Number analyzed (Participants) | 992 | 829 | 1150 | 2971
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (16.0) | 50.9 (16.0) | 52.6 (16.0) | 51.7 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 590 | 514 | 688 | 1792
  Male | 402 | 315 | 462 | 1179
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 108 | 131 | 112 | 351
  Not Hispanic or Latino | 884 | 698 | 1038 | 2620
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 4 | 7 | 17
  Asian | 18 | 17 | 38 | 73
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 202 | 77 | 115 | 394
  White | 640 | 598 | 860 | 2098
  More than one race | 13 | 6 | 13 | 32
  Unknown or Not Reported | 113 | 127 | 117 | 357

OUTCOME MEASURES:

1. Primary Outcome: Spine-related Cost of Care at One Year
Description: Measured by patient self-report
Time Frame: One year
Population: The primary analytic cohort included patients who consented AND completed baseline questionnaires.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Usual PCP Led Care | Identify, Coordinated, Enhanced (ICE) Decision Making | Individualized Postural Therapy (IPT)
Number analyzed (Participants) | 992 | 829 | 1150
dollars | 1587 (5774) | 1448 (2756) | 2528 (2756)
Statistical Analysis 1: Comparison: Usual PCP Led Care vs Identify, Coordinated, Enhanced (ICE) Decision Making; Test type: Superiority; p = .04, GEE with log link and Poisson errors; Risk Ratio (RR) = .93, 95% CI 2-sided [.87 to .997]
Statistical Analysis 2: Comparison: Usual PCP Led Care vs Individualized Postural Therapy (IPT); Test type: Superiority; p < 0.001, GEE with log link and Poisson errors; Risk Ratio (RR) = 1.40, 95% CI 2-sided [1.35 to 1.45]

2. Primary Outcome: Change in Pain
Description: Measured by Oswestry Disability Index The Oswestry Disability Index (ODI) captures pain related disability based on patient self-report.
  The ODI ranges from 0 (best) to 100 (worst). The Minimal clinically important difference (MCID) for ODI in patients with spine pain is 6 points.
  The change in participant-level pain related disability from baseline to 3 months using the Oswestry Disability Index has been reported.
  Reference: Fairbank JCT, Couper J, Davies JB, O'Brien JP. The Oswestry Low Back Pain Disability Questionnaire. Physiotherapy. 1980;66:271-273
Time Frame: Three months
Population: The analytic cohort included patients who consented AND completed baseline questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual PCP Led Care | Identify, Coordinated, Enhanced (ICE) Decision Making | Individualized Postural Therapy (IPT)
Number analyzed (Participants) | 992 | 829 | 1150
score on a scale | -9.4 (18.3) | -15.9 (16.2) | -13.9 (15.9)
Statistical Analysis 1: Comparison: Usual PCP Led Care vs Identify, Coordinated, Enhanced (ICE) Decision Making; Test type: Superiority; p < 0.001, GEE with identity link and normal errors; Risk Difference (RD) = -5.8, 95% CI 2-sided [-7.7 to -3.9]
Statistical Analysis 2: Comparison: Usual PCP Led Care vs Individualized Postural Therapy (IPT); Test type: Superiority; p < 0.001, GEE with identity link and normal errors; Risk Difference (RD) = -4.3, 95% CI 2-sided [-5.9 to -2.6]

3. Secondary Outcome: Change in Pain
Description: Measured by Oswestry Disability Index The Oswestry Disability Index (ODI) captures pain related disability based on patient self-report.
  The ODI ranges from 0 (best) to 100 (worst). The MCID for ODI in patients with spine pain is 6 points.
  The change in participant-level pain related disability from baseline to 12 months using the Oswestry Disability Index has been reported.
  Reference: Fairbank JCT, Couper J, Davies JB, O'Brien JP. The Oswestry Low Back Pain Disability Questionnaire. Physiotherapy. 1980;66:271-273
Time Frame: One year
Population: The analytic cohort included patients who consented AND completed baseline questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual PCP Led Care | Identify, Coordinated, Enhanced (ICE) Decision Making | Individualized Postural Therapy (IPT)
Number analyzed (Participants) | 992 | 829 | 1150
score on a scale | -9.2 (18.9) | -17.7 (16.4) | -16.3 (16.1)
Statistical Analysis 1: Comparison: Usual PCP Led Care vs Identify, Coordinated, Enhanced (ICE) Decision Making; Test type: Superiority; p < 0.001, GEE with identity link and normal errors; Risk Difference (RD) = -7.5, 95% CI 2-sided [-9.4 to -5.7]
Statistical Analysis 2: Comparison: Usual PCP Led Care vs Individualized Postural Therapy (IPT); Test type: Superiority; p < 0.001, GEE with identity link and normal errors; Risk Difference (RD) = -6.7, 95% CI 2-sided [-8.4 to -5.0]

4. Secondary Outcome: Quality of Life (EQ5D-5L VAS Scores)
Description: EuroQol 5-Dimensional Visual Analogue Scale (EQ-5D-5L VAS) by the EuroQol Group measures patient's self-rated health-related quality of life on a vertical visual analog scale.
  EQ-5D-5L VAS range from 0 to 100, with 100 indicating the best score. The MCID for the EQ-5D-5L visual analogue scale ranges from 5.3 to 10.5.
  The health-related quality of life at 12 months using the EQ-5D-5L VAS has been reported.
Time Frame: One year
Population: The analytic cohort included patients who consented AND completed baseline questionnaires.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Usual PCP Led Care | Identify, Coordinated, Enhanced (ICE) Decision Making | Individualized Postural Therapy (IPT)
Number analyzed (Participants) | 992 | 829 | 1150
score on a scale | 3.2 [1.8 to 4.5] | 8.9 [7.7 to 10.2] | 10.5 [9.4 to 11.6]
Statistical Analysis 1: Comparison: Usual PCP Led Care vs Identify, Coordinated, Enhanced (ICE) Decision Making; Test type: Superiority; p < 0.001, GEE with identity link and normal errors; Risk Difference (RD) = 4.7, 95% CI 2-sided [2.6 to 6.8]
Statistical Analysis 2: Comparison: Usual PCP Led Care vs Individualized Postural Therapy (IPT); Test type: Superiority; p < 0.001, GEE with identity link and normal errors; Risk Difference (RD) = 6.0, 95% CI 2-sided [4.1 to 7.9]

5. Secondary Outcome: Self-efficacy
Description: The Lorig self-efficacy functioning sub-scale items ask individuals how confident they are in performing certain daily activities.
  Lorig self-efficacy functioning sub-scale scores range from 0 to 100, with 100 indicating the best score. The MCID for the Lorig self-efficacy scale has not been established.
  The patient-reported self-efficacy at 12 months using the Lorig self-efficacy functioning sub-scale has been reported.
  Reference: Lorig K, Chastain RL, Ung E, Shoor S, Holman HR. Development and evaluation of a scale to measure perceived self-efficacy in people with arthritis. Arthritis Rheum. 1989 Jan;32(1):37-44. doi: 10.1002/anr.1780320107. PMID: 2912463.
Time Frame: One year
Population: The analytic cohort included patients who consented AND completed baseline questionnaires.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Usual PCP Led Care | Identify, Coordinated, Enhanced (ICE) Decision Making | Individualized Postural Therapy (IPT)
Number analyzed (Participants) | 992 | 829 | 1150
score on a scale | -1.0 [-2.3 to .3] | 7.4 [6.4 to 8.4] | 6.4 [5.4 to 7.3]
Statistical Analysis 1: Comparison: Usual PCP Led Care vs Identify, Coordinated, Enhanced (ICE) Decision Making; Test type: Superiority; p < 0.001, GEE with identity link and normal errors; Risk Difference (RD) = 6.8, 95% CI 2-sided [5.0 to 8.7]
Statistical Analysis 2: Comparison: Usual PCP Led Care vs Individualized Postural Therapy (IPT); Test type: Superiority; p < 0.001, GEE with identity link and normal errors; Risk Difference (RD) = 6.7, 95% CI 2-sided [5.0 to 8.4]

ADVERSE EVENTS:
Description: Adverse events were not assessed
Arm/Group | Usual PCP Led Care | Identify, Coordinated, Enhanced (ICE) Decision Making | Individualized Postural Therapy (IPT)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT03083886/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT03083886/ICF_001.pdf